CLINICAL TRIAL: NCT02501278
Title: A Phase II Clinical Trial of Chemo-radiotherapy in Combination With INO-3112 in Patients With Locally Advanced Cervical Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: company (Inovio) is no longer able to support the study
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Collaborators: Inovio Pharmaceuticals (Industry); Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-1411; 2015-004602-42 (EudraCT Number)
Record Dates: First submitted 2015-07-07; First posted 2015-07-17 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Uterine Cervical Neoplasms
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — MEDI0457; Radiotherapy; Brachytherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm A: Immunotherapy during and after CRT + vaccine boost (Experimental): INO-3112 dosing during chemoradiotherapy plus immunotherapy dosing after chemoradiotherapy in an adjuvant setting and vaccine boost one year after last vaccine dosing.
  Interventions: Biological: INO-3112 vaccine; Radiation: Radiotherapy (Extrernal beam radiotherapy + brachytherapy); Drug: Cisplatin chemotherapy
- Arm B: Immunotherapy during CRT + vaccine boost (Experimental): INO-3112 dosing during chemoradiotherapy, and vaccine boost one year after last vaccine dosing.
  Interventions: Biological: INO-3112 vaccine; Radiation: Radiotherapy (Extrernal beam radiotherapy + brachytherapy); Drug: Cisplatin chemotherapy
- CRT without immunotherapy (Active Comparator): Standard chemoradiotherapy without immunotherapy
  Interventions: Radiation: Radiotherapy (Extrernal beam radiotherapy + brachytherapy); Drug: Cisplatin chemotherapy

INTERVENTIONS:
Biological: INO-3112 vaccine — INO-3112 i.e. the combination of VGX-3100 and INO-9012, specifically:
  * VGX-3100 (HPV16 and HPV18 E6-E7 DNA vaccine) will be administered at 3 mg per plasmid (6 mg total DNA)
  * INO-9012 (IL-12 DNA plasmid) will be administered at 1 mg per dose will be administered using the CELLECTRA® electoporation device
  Arms: Arm A: Immunotherapy during and after CRT + vaccine boost; Arm B: Immunotherapy during CRT + vaccine boost
Radiation: Radiotherapy (Extrernal beam radiotherapy + brachytherapy) — The whole pelvis will be irradiated with 45 - 50.4 Gy in 25-28 fractions in fractions of 1.8 Gy over 5 weeks daily.
  Those patients with pelvis positive and/or para-aortic positive lymph nodes should be treated with an elective dose to the para-aortic area of 45 Gy in fractions of 1.6-1.8 Gy in 25-28 fractions.
  Pelvic and para-aortic nodes known to contain gross/macroscopically visible disease and heavily involved parametria or tumor areas that may lie beyond the high-dose range of brachytherapy should be treated with additional small volume boost of EBRT to a total dose of 60-65 Gy using a combination of either sequential and/or concomitant boost. Fractions of 1.8-2 Gy can be used in the sequential boost.
Drug: Cisplatin chemotherapy — Cisplatin chemotherapy will be administered i.v. at a dose of 40 mg/m2 (total 5 cycles during week 1-5) weekly in concomitance with RT with the total dose not to exceed 70 mg per week.

SUMMARY:
The aim of this study is to assess the potential benefit of the addition of immunotherapy with VGX-3100 and INO-9012 (i.e. INO-3112) to concomitant CRT or, to concomitant CRT and continued as adjuvant in patients with locally advanced cervical cancer.

Safety run-in: To test the safety of CRT combined with immunotherapy with INO-3112. This safety run-in phase will include the first 3 patients treated in each of the two INO-3112 combination arms who are exposed to at least two immunotherapy doses and evaluate whether the combination does not pose undue immediate risks to the patients further enrolled in the trial.

Phase II:To demonstrate sufficient activity in the experimental combination arms to warrant a further phase III conclusive trial based on progression free survival (PFS) at 18 months assessed by RECIST by the local investigator. The efficacy will be assessed within each experimental arm while the standard arm will serve as a reference arm to check the reliability of the results.

ELIGIBILITY:
Main inclusion criteria:

Registration step

* Age 18 years or older;
* Newly diagnosed locally advanced cervical cancer defined as FIGO 2009: stage IB2, IIA&IIB, IIIA&IIIB or IVA disease;
* No evidence of distant metastases (Stage IVB);
* Histological diagnosis of squamous cell carcinoma, adenocarcinoma or adenosquamous cell carcinoma of the cervix is accepted. Not accepted are small cell, clear cell and other rare variants of the classical adenocarcinoma;
* Availability of HPV 16 and HPV 18 testing;
* No HIV seropositive, Hepatitis B or C (unless sustained virologic response achieved by anti-HCV therapy);
* Written informed consent must be given according to ICH/GCP, and national/local regulations

Randomization step

* Positive for HPV 16 and/or HPV 18 as assessed by central lab;
* WHO/ECOG performance status 0 - 2
* Adequate hematological, liver and renal functions
* ECG with no clinically significant findings as assessed by the investigator performed within 30 days of signing the informed consent form
* Absence of current malignancies at other sites, with the exception of adequately treated basal or squamous cell carcinoma of the skin. Cancer survivors, who have undergone potentially curative therapy for a prior malignancy, who have no evidence of that disease for five years and are deemed at low risk for recurrence, are eligible for the study;
* No prior history of clinically significant autoimmune disease, Crohn's disease, ulcerative colitis;
* No history of previous therapeutic HPV vaccination (individuals who have been immunized with licensed prophylactic HPV vaccines (e.g. Silgard®, Cervarix®, Gardasil®) are not excluded);
* No known or suspected hypersensitivity to component(s) of investigational product or cisplatin contraindication (e.g. peripheral neuropathy ≤ grade 2 or ototoxicity ≤ grade 2 as per CTCAE v4);
* No previous pelvic RT;
* No previous chemotherapy for this tumor;
* No patients who have undergone a previous hysterectomy or will have a hysterectomy as part of their initial cervical cancer therapy;
* No receipt of any immunotherapy within 4 weeks of start of protocol treatment;
* No prior major surgery within 4 weeks of randomization from which the patient has not recovered.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-05; Primary Completion 2019-05 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Occurence of Adverse Events | 6 months
  In order to ensure adequate safety of the combination treatment, a safety run-in will be performed. This safety run-in phase will include the first 3 patients treated in each of the experimental arms (arms A & B) exposed to at least two immunotherapy doses. The acute safety of the combination of INO-3112 with concomitant CRT will be evaluated similar to a phase I "3+3" safety design. The safety evaluation will be done by the Data Safety Monitoring Board who will invoke an IDMC evaluation of the whole study if undue safety signals are observed.
  Acute toxicity is defined as a grade 3 or more related AEs occurring between the first dose of vaccine administration and up to 14 days after the second dose of immunotherapy. Adverse events are graded according to the NCI CTCAE v4.0. Use of narcotics will be reviewed on case-to-case basis by a medical review team to assess its relevance towards the safety evaluation
Progression free survival (PFS) at 18 months assessed by RECIST | 18 months
  Progression Free Survival at 18 months assessed by local investigator

CONTACTS AND LOCATIONS:
Overall Officials: Fernanda Herrera, Study Chair — Centre hospitalier universitaire vaudois, Lausanne; George Coukos, Study Chair — Centre hospitalier universitaire vaudois, Lausanne
Locations (1):
- Centre Hospitalier Universitaire Vaudois, Lausanne, Switzerland